CLINICAL TRIAL: NCT00229775
Title: Efficacy of Chloroquine + Sulfadoxine Pyrimethamine Versus Artemether + Lumefantrine for the Treatment of Uncomplicated Plasmodium Falciparum Malaria in the Philippines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Department of Health, Philippines (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCID-3913; U30/CCU317876-01
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Malaria
Keywords: Plasmodium falciparum malaria; malaria; artemether lumafantrine; chloroquine; sulfadoxine pyrimethamine; Coartem
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Artemether

INTERVENTIONS:
Drug: artemether/lumafantrine vs chloroquine/sulfadoxine-pyrimethamine

SUMMARY:
The purpose of this study is to determine whether artemether + lumefantrine is as effective as chloroquine + sulfadoxine pyrimethamine in the treatment of uncomplicated Plasmodium falciparum malaria

DETAILED DESCRIPTION:
Background: In the Philippines, close to 11 million people in 65 provinces are at risk for acquiring malaria infections. It is still one of the ten leading causes of morbidity nationwide. Each day, roughly 150-200 people fall ill with malaria. In the past 40 years, the mortality rate stabilized at around 2/100,000 population. Of those people who have malaria, approximately 1% die per year. Malaria remains one of the major causes of death in provinces such as Palawan, Isabela, Tawi-tawi, Sulu and Butuan City. Approximately 70% of all malaria in the Philippines is Plasmodium falciparum with the remaining species being P. vivax.

Recently the Department of Health (DOH) instituted a change in the national antimalarial drug guidelines changing from using chloroquine (CQ) and sulfadoxine pyrimethamine (SP) monotherapy as first and second line drugs, respectively, to a combined chloroquine plus sulfadoxine-pyrimethamine as first-line treatment, and artemether-lumefantrine (Coartem) as second line treatment. This change was made due to increasing levels of drug resistance to the previous first and second-line therapies. In order to have an improved understanding of the trends of antimalarial drug resistance in the Philippines, the DOH is initiating a sentinel surveillance system for monitoring of antimalarial drug resistance. Three sites have been selected to be representative of the country.

Objective: To establish a sentinel surveillance system to assess the efficacy of chloroquine plus sulfadoxine-pyrimethamine versus artemether + lumefantrine for the treatment of uncomplicated P. falciparum infections in three areas of the Republic of the Philippines.

Methods: An in vivo antimalarial drug efficacy trial will be conducted in three areas of the Philippines. Subjects > 6 months of age with parasitologically confirmed, uncomplicated P. falciparum infections will be recruited. Patients will be treated with single dose SP (25 mg/kg of the sulfadoxine component in a single dose) plus CQ (25 mg/kg over three days) or artemether + lumefantrine (twice daily) over 3 days. Patients will be randomly assigned one of the two drugs regimens. Clinical and parasitological parameters will be monitored over a 28-day follow-up period to evaluate drug efficacy. Results from this study will be used to assist the DOH in assessing their national malaria treatment policy for P. falciparum malaria.

ELIGIBILITY:
Inclusion Criteria:

1. Weight > 10 kg;
2. Documented fever (axillary temperature >37.5oC) and/or a history of fever during the previous 24 hours in the absence of another obvious cause of fever (such as pneumonia, measles, otitis media);
3. Monoinfection with P. falciparum between 1,000 and 100,000 asexual parasites/µl as determined by microscopic examination of thick, or thick and thin peripheral blood smears;
4. Informed consent from the patient or parent/guardian (in the case of children),assent from child (ages 8 -17 years inclusive);
5. Willingness on the part of the patient to return to the clinic for regular check-ups during the 28-day follow-up period.

Exclusion Criteria:

1. Danger signs: unable to drink or breastfeed; vomiting (more than twice in the previous 24 hours); recent history of convulsions (one or more in the previous 24 hours); impaired consciousness; unable to sit or stand; 2. Severe Manifestations of P. falciparum malaria in adults and children (World Health Organization criteria)

1. Prostration (inability to sit unassisted [children], extreme weakness [adults])
2. Impaired consciousness (Blantyre coma scale [children], Glascow coma scale [adults])
3. Respiratory distress (sustained nasal flaring, indrawing, Kussmaul breathing)
4. Multiple convulsions (³2 convulsions/24 hour period)
5. Circulatory collapse (hypotension and poor perfusion)
6. Pulmonary edema
7. Abnormal bleeding
8. Jaundice
9. Hemoglobinuria
10. Severe anemia (Hb < 5 gm/dL)
11. Hypoglycemia (blood glucose < 2.2 mmol/L [<40 mg/dL])
12. Acidosis (bicarbonate <15 mmol/L)
13. Hyperparisitemia (level varies with endemicity)
14. Renal impairment (urine output < 12 mL/kg/24 hours) 3. Other underlying chronic or severe diseases (e.g., cardiac, renal, hepatic diseases, HIV/AIDS, malnutrition); 4. History of hypersensitivity reactions to any of the drugs being tested or used as alternative treatment: sulfonamides, chloroquine, artemisinins, artemether, lumefantrine, quinine or tetracycline/clindamycin; 4. Pregnancy (history of pregnancy or a positive urine pregnancy test); 5. Women who are breast feeding children less than 8 weeks of age. -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2003-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Clinical cure

SECONDARY OUTCOMES:
Hemoglobin levels

CONTACTS AND LOCATIONS:
Overall Officials: Dorin Bustos, MD, PhD, Study Director — RITM, DOH, Philippines
Locations (3):
- Philippines (3):
  - Kalinga Health Center, Tabuk, Kalinga Province
  - Davao Health Center, Davao City, Mindinao
  - Palawan Health Center, Puerto Princesa City, Palawan